CLINICAL TRIAL: NCT02729103
Title: Treatment Patterns, Mortality, Healthcare Resource Utilization, and Costs in Patients With Prostate Cancer With Bone Metastases: A Retrospective Database Analysis .
Brief Title: Treatment Patterns in Metastatic Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18695
Record Dates: First submitted 2016-03-16; First posted 2016-04-06 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment patterns, healthcare resource utilization and costs: Part 1 - Assessment of treatment patterns, healthcare resource utilization and costs. The study cohort will include all patients with prostate cancer with incident bone metastases during the index period (1 June 2013 to 1 July 2014) based on a large database encompassing a broad sample of the commercially insured U.S. population. The first date of bone metastases diagnosis or first date of treatment indicative of bone metastases (whichever occurs first) will be designated as the index date. All patients must have no diagnosis of other cancers, no diagnosis of bone metastases or a claim for a treatment indicative of bone metastases, and no skeletal-related events (SREs) in the 12-month pre-index period. Additionally, all subjects must be continuously enrolled for at least 12 months before and at least 6 months after the index date.
  Interventions: Drug: Xofigo (Radium 223 dichloride,BAY88-8223)
- Mortality: Part 2 - Assessment of mortality. The study cohort will include all patients with prostate cancer with incident bone metastases during the index period (1 June 2013 to 1 July 2014) based on a large database encompassing a broad sample of the commercially insured U.S. population. The first date of bone metastases diagnosis or first date of treatment indicative of bone metastases (whichever occurs first) will be designated as the index date. All patients must have no diagnosis of other cancers, no diagnosis of bone metastases or a claim for a treatment indicative of bone metastases, and no SREs in the 12-month pre-index period. Additionally, all subjects must be continuously enrolled for at least 12 months before the index date. Unlike in Part 1, there will be no required minimum follow-up time after the index date (in order to assess mortality).
  Interventions: Drug: Xofigo (Radium 223 dichloride,BAY88-8223)

INTERVENTIONS:
Drug: Xofigo (Radium 223 dichloride,BAY88-8223) — Retrospective claims analysis. Descriptive analyses of treatment patterns.

SUMMARY:
This study will evaluate treatment patterns, mortality, healthcare resource utilization, and costs in patients with prostate cancer with bone metastases (primary objectives). Additionally, this study will evaluate opioid/analgesic use among lines of therapy in this patient population (secondary objective). The study is descriptive in nature and is meant to provide a greater understanding of the patterns of therapy observed in real-world clinical practice (in the absence of clear guideline recommendations with regards to treatment sequencing), to contribute to a greater understanding of the major cost drivers (thus better-informing payers), and to examine real-world mortality in such patients.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with at least one claim with a primary diagnosis of prostate cancer (International Classification of Diseases(ICD) Clinical Modification (CM)185.xx )and any of the below on same day or after the prostate cancer claim:

* At least one inpatient claim with a primary or secondary diagnosis indicating bone metastases (ICD 9 CM 198.5 or Healthcare Common Procedure Coding System (HCPCS) code for a treatment indicative of bone metastases OR
* At least two outpatient claims with a primary or secondary diagnosis indicating bone metastases (ICD 9 CM 198.5 or HCPCS code for a treatment indicative of bone metastases, with a minimum of 30 days between claims.

Exclusion Criteria:

* Subjects with a diagnosis of a cancer other than prostate cancer - defined as the presence of one inpatient or two outpatient claims with a primary or secondary diagnosis of malignant neoplasms (ICD-9-CM 140.xx-171.xx, 174.xx-184.xx,186.xx-195.xx,200.xx-209.3x, 230.xx-239.xx) - in the 12-month pre-index period.
* Subjects with any claim for a primary or secondary diagnosis indicating bone metastases (ICD-9-CM 198.5) or any treatment indicative of bone metastases in the 12-month pre-index period.
* Patients who had a SRE in the 12-month pre-index period.
* Subjects without continuous enrollment for at least 12 months before the index date.
* Subjects without continuous eligibility for at least 6 months after the index date.
* Subjects that are female.
* Subjects that have negative costs.
* Subjects that are less than 45 years of age on the index date.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1 - Assessment of treatment patterns, healthcare resource utilization, and costs The study cohort will include all patients with prostate cancer with incident bone metastases during the index period (1 June 2013 to 1 July 2014) based on a large database encompassing a broad sample of the commercially insured U.S. population. The first date of bone metastases diagnosis or first date of treatment indicative of bone metastases (whichever occurs first) will be designated as the index date.
  Part 2 - Assessment of mortality The study cohort will include all patients with prostate cancer with incident bone metastases during the index period (1 June 2013 to 1 July 2014) based on a large database encompassing a broad sample of the commercially insured U.S. population. The first date of bone metastases diagnosis or first date of treatment indicative of bone metastases (whichever occurs first) will be designated as the index date.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Distribution of treatment types among lines of therapy | Up to 6 months
  Possible Treatment Types: Sipuleucel-T, Abiraterone, Enzalutamide, Docetaxel, Cabazitaxel, Radium-223, Anti-Androgens, All other chemotherapy(oral and injectables), Radiation therapy
Time to treatment (days) | Up to 6 months
Duration of treatment (days) | Up to 6 months
Number of patients on each drug or drug combination | Up to 6 months
  Drug: Sipuleucel-T, Abiraterone, Enzalutamide, Docetaxel, Cabazitaxel, Radium-223, Anti-Androgens, All other chemotherapy(oral and injectables), Radiation therapy
Number of inpatient visits per patient | Upto 6 month post index period
Length of hospital stay (days) among those with an inpatient visit | Upto 6 month post index period
Number of outpatient visits per patient | Upto 6 month post index period
Number of emergency room (ER) visits per patient | Upto 6 month post index period
Number of physician office visits per patient | Upto 6 month post index period
Number of medication prescriptions per patient | Upto 6 month post index period
Number of patients by provider type | Upto 6 month post index period
Number of claims per patient | Upto 6 month post index period
Total costs of healthcare | Upto 6 month post index period
Medical costs of healthcare | Upto 6 month post index period
Pharmacy costs of healthcare | Upto 6 month post index period
Per-patient-per-month (PPPM)) costs of healthcare | Upto 6 month post index period
Mortality rate | Up to 6 months

SECONDARY OUTCOMES:
Opioid/analgesic use among lines of therapy(Y/N) | Up to 6 months
  Opioid and analgesics use among lines of therapy (e.g. 1st, 2nd, 3rd)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Whippany, New Jersey, United States